CLINICAL TRIAL: NCT03966248
Title: Chinese Tuina (Chinese Massage and Manipulation Therapy) for KOA: A Randomized, Parallel, Physical Therapies Active Controlled Study
Brief Title: Chinese Tuina Therapy for Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Changhe Yu, Principal Investigator, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DZM-KY201906
Record Dates: First submitted 2019-05-26; First posted 2019-05-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthritis; Massage; Tuina; Traditional Chinese medicine; Physical therapy; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; manual therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: Two arms recruit and evaluate the participants at the same time, and the included participants have the equal opportunity to either the Chinese Tuina or physical manual therapy groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are randomly divided into Chinese Tuina group and Physical Manual group at a ratio of 1:1, only knowing that they will receive the manual therapies. The assessor, data manager and statistician will not participate in the randomized process and the treatment and share any information with each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese Tuina group (CTG) (Experimental): The participants in CT group will receive the traditional Chinese Tuina therapy on the basis of KOA health education and home-exercise.
  Interventions: Other: Chinese Tuina therapy
- Physical Manual group (PMG) (Active Comparator): The participants in PM group will receive the modern physical manual therapy on the basis of KOA health education and home-exercise.
  Interventions: Other: Physical Manual therapy

INTERVENTIONS:
Other: Chinese Tuina therapy — 1. The doctor presses the affected lower limb from the anterior superior iliac spine to the ankle;
  2. The doctor gives the pressure on the Biguan(ST31), Futu(ST32), Heding(EX-LE2), Neixiyan(EX-LE4), Waixiyan(Dubi, ST35), Zusanli(ST36) and Sanyinjiao(SP6) of the affected lower limb;
  3. Massage the spleen and stomach meridians of the affected lower extremes;
  4. Roll the soft tissues around the affected knee;
  5. Relax the gastrocnalis muscle
  6. The doctor gives the pressure on the Xuehai(SP10), Liangqiu(ST34), Neixifeng(medial patellofemoral ligament), Waixifeng(lateral patellofemoral ligament), Neixiyan(EX-LE4) and Waixiyan(Dubi, ST35) at the same time;
  7. Push the patella and do the passive movement of the affected knee;
  8. Strength training of the affected knee.
  This group receives 8 treatments over a 3 week period with a one week follow-up on site and a 3 month follow-up by mail, phone or email.
  Arms: Chinese Tuina group (CTG)
Other: Physical Manual therapy — 1. Manual therapy: Stretching the knee joint, stretching the knee joint with valgus or abduction, stretching the knee joint with varus or adduction is suitable for patients with knee flexion and extension difficulty.Patellar manipulation by bending the knee 5-10 degrees downward is suitable for patients with patellar sliding difficulty.The lower end of the muscle length manipulation is suitable for patients with muscle tension and soft tissue tension.Soft tissue loosening is performed in the suprapatellar and peripatellar regions, medial and lateral capsule joints, and popliteal fossa.
  2. Activity training: Mainly about the knee joint flexion and extension movement training.
  3. Strength training: Mainly about quadriceps muscle resistance exercises
  This group receives 8 treatments over a 3 week period with a one week follow-up on site and a 3 month follow-up by mail, phone or email.
  Arms: Physical Manual group (PMG)

SUMMARY:
Knee osteoarthritis (KOA) is one of the most common musculoskeletal diseases in clinic. It usually occurs in middle-aged people, especially women. An estimated lifetime risk for KOA is approximately 40% in men and 47% in women. KOA is a chronic disease which can lead to obvious pain, joint stiffness, limitation of activity and even disability, with significant associated costs and effects on society, health systems, and individuals. Tuina therapy has been used and showed effectiveness and safety for pain relief and disability for the patients with musculoskeletal disorders for years in China. Though it is regarded that the Traditional Chinese medicine (TCM) Tuina therapy is similar to the modern manual therapies, the modalities of TCM tuina therapy are different and effect maybe equal to or more better than the modern manual therapy in clinic. However, little evidence exists that Tuina benefits the KOA. The investigators will do this in a randomized, parallel, active controlled study to observe whether TCM Tuina is more beneficial to KOA than the physical manual therapy, which has been considered an effective and standard care for KOA.

DETAILED DESCRIPTION:
Patients will be randomly allocated to one of two groups. In the Chinese Tuina group (group CTG), patients will receive the traditional Chinese Tuina therapy (including rolling, grasping, scratching, pressing, acupressure or pushing) on the basis of KOA health education and home-exercise. Patients in the Physical Manual group (group PMG) will receive the modern physical manual therapy (including joint mobilization/manipulation, manual traction, soft tissue manipulations, passive stretching, range of motion and strength training) on the basis of KOA health education and home-exercise. Assessments will be conducted at baseline and 4 and 16 weeks after randomization.

It is expected that the interventions will alleviate the sufferings of the patient. The risks of participation are minimal. Occasionally, tuina can make people feel nauseous or experience a temporary increase in pain either during or after treatment. Rare side effects happen during and after Tuina or manual treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of KOA;
2. Age 40-75 years;
3. KL (Kellgren-Lawrence) grade Ⅱ or Ⅲ in recent 3 months;
4. NRS score of pain at least more than 4 points;
5. Single/bilateral knee pain, duration of more than 6 month; If the patient has KOA on both legs, the heavier leg is selected for study.

Exclusion Criteria:

1. Surgery history of knee or waiting for surgery (knee replacement or knee arthroscopy);
2. Knee pain caused by other diseases (such as joint bodies, severe effusion of joint cavity, infection, malignant tumors, autoimmune diseases, trauma, etc.);
3. Oral administration of hormones within 3 month, intra-articular injection within 6 months, knee injuries or open injuries within 6 months, or knee arthroscopy within 1 year.
4. Severe acute/chronic organic or mental diseases;
5. Pregnant women, pregnant and lactating women;
6. Coagulation disorders (such as hemophilia, etc.), or the skin diseases at the site of operation;
7. Device support treatment after knee osteoarthritis disability;
8. Participation in another clinical study in the past 3 months;
9. History of receiving acupuncture, massage, manipulation, or any medical plaster treatment within 3 months
10. Breaks for treatment longer than 3-4 weeks depending on each circumstance or merit may be construed as non-compliance and may be excluded.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Change from baseline at 4 weeks
  Self report measure of pain, stiffness, and physical function for people with knee osteoarthritis.

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Change from baseline at 8 weeks and 16 weeks
  Self report measure of pain, stiffness, and physical function for people with knee osteoarthritis.
Change in Numeric Knee Pain Rating Scale | Change from baseline at 4 weeks, 8 weeks and 16 weeks
  Subjects will rate their worst knee pain in the last 24 hours using an 11 point numeric pain rating scale with 0 representing "no pain" and 10 representing " the worst pain imaginable".
Change in Patient Global Assessment (PGA) | Change from baseline at 4 weeks, 8 weeks and 16 weeks
  The Patient global assessment rating is a 11 point Numeric Rating Scale in which subjects will rate the degree to which their knee condition has changed from the time treatment was initiated to the present. The subject responds to the following query: "Please rate your overall knee's condition from the time you began treatment until now." using an 11 point numeric rating scale with 0 representing "A very great deal better" and 10 representing "A very great deal worse".
Change in 12-item Short Form Health Survey (SF-12) | Change from baseline at 4 weeks, 8 weeks and 16 weeks
  The SF-12 is a generic health-related quality of life measure.
Change in 30 second time chair rise test | Change from baseline at 4 weeks
  Subjects will be seated with their arms crossed in front of their chest. On the command "go" subjects will stand up and sit down for as many trials as they can in a 30 second period.
Change in Timed Up and Go Test Time | Change from baseline at 4 weeks
  On the command "go" subjects will stand up from a chair, walk 3 meters, turn around, return to the chair and sit down. The time it takes to complete this task will be recorded.
Change in One Leg Standing Test | Change from baseline at 4 weeks
  One single-leg standing was assessed balance. Test required the subject to stand with arms by his/her side.Timing was started when the subject raised one foot off the ground. Timing was stopped if the subject displaced the weight-bearing foot, touched the suspended foot to the ground, used the suspended limb to support the weight-bearing limb, or reached the maximum balance time of 30 seconds.
OARSI Responder Criteria | At weeks 4 after randomisation.
  Responder criteria included 1) greater than or equal to 50% improvement in WOMAC pain or WOMAC function and an absolute improvement of greater than or equal to 20, or 2) improvement in at least 2 of the following 3 scores: 20% improvement in pain and absolute change ≥ 10 on WOMAC pain score, 20% improvement in pain and absolute change ≥ 10 on WOMAC function score, or moderate or greater improvement (≤ 4) on a 15 point global rating of change scale
Blinding assessment | At weeks 4 after randomisation.
  To test whether the participants are blinded successfully, all participants will be asked to guess which kind of treatment they received.
Credibility/Expectancy Questionnaire | About 5 min after the first treatment
  The credibility and expectancy of participants will be measured using the Credibility/Expectancy Questionnaire
Rescue medicine | At weeks 4, 8 and 16 after randomisation.
  Any use of pain-killers will be ascertained.
Adverse events | At weeks 4 after randomisation.
  Adverse Event Form

CONTACTS AND LOCATIONS:
Overall Officials: Xiyou Wang, Principal Investigator — Beijing University of Chinese Medicine affiliated Dongzhimen Hospital
Locations (1):
- Dongzhimen hospital affiliated to Bejing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma P, Liu L, Li S, Cai M, Han S, Weng Z, Chen Q, Gao Y, Zhang L, Wu G, Yang X, Zhang Y, Li D, Liu C, Sun Y, Yan S, Wang X, Yu C. Comparative effectiveness of Tuina therapy versus manual physical therapy for knee osteoarthritis: a randomized controlled trial. BMC Complement Med Ther. 2025 Apr 8;25(1):128. doi: 10.1186/s12906-025-04850-w. PMID 40200237